CLINICAL TRIAL: NCT06715787
Title: Evaluating the Food Education Access Support Together (FEAST) Perinatal Support Program: A Randomized Controlled Trial
Brief Title: FEAST Perinatal Support Program Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Tyler Mason, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APP-24-02282; P50MD017344 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-12-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Diet, Healthy; Obesity; Cardiometabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: One treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FEAST Perinatal Support Program (Experimental): Active behavioral intervention
  Interventions: Behavioral: FEAST Perinatal Support Program

INTERVENTIONS:
Behavioral: FEAST Perinatal Support Program — The intervention will include the core perinatal support program (PSP) with $15 weekly grocery gift cards for healthful food (fruit, vegetables, whole grains), The PSP will be completed during weekly group sessions over 16 weeks. The core PSP includes the two primary behavior change techniques: group-based nutrition education based on current United States Department of Agriculture (USDA) national guidelines for pregnant individuals and guided group sharing and engagement.

SUMMARY:
Latino individuals face an elevated risk of adverse health outcomes during pregnancy, impacting both the birthing parent and the baby with potential long-term chronic health conditions. While promoting a healthy diet during pregnancy is a promising strategy, interventions targeting dietary behaviors have yielded mixed results and lack widespread dissemination in communities in need. Collaborating with community-based organizations could enhance cultural relevance, build trust with Latino families, and improve program reach and effectiveness. Food Education Access Support Together (FEAST) is a community-based program that promotes healthy eating, well-being, and health equity for diverse, under-resourced urban populations in Los Angeles. The newly developed FEAST Perinatal Support Program (PSP) aims to support individuals through pregnancy and postpartum by providing dietary psychoeducation, skill-building, and social support, with an additional component of grocery gift cards to address food access barriers. This study proposes a pilot trial to assess the feasibility and preliminary efficacy of the FEAST PSP in enhancing dietary outcomes, overall health, and socio-cognitive precursors, in pregnant individuals. The study will enroll 40 pregnant adults in a single-arm study who will receive the core PSP with a $15 gift card for healthful fresh food (PSP+giftcard). Pre- and post-intervention assessments will include questionnaires, dietary recalls, physical measurements, and interviews to evaluate program perceptions. Specific aims include evaluating program feasibility and acceptability (i.e., reach, retention, and participant perceptions) and determining preliminary efficacy on changing socio-cognitive and behavioral aspects of diet, self-reported health, and cardiometabolic risk factors. The project aligns with goals of improving health outcomes in Latino families in Southern California and supports FEAST's strategic objectives for improving health and wellness of individuals during pregnancy and throughout the lifespan. The findings will inform program refinement and future NIH grants for rigorous evaluation of the FEAST PSP.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* Speak and read English
* Eligible for Electronics Benefit Transfer (EBT) and/or Women, Infants, and Children (WIC) benefits

Exclusion Criteria:

* Inability to attend in-person sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mini-EAT 9-item score | Survey at baseline and immediately post-assessment
  Aggregate score of 9 items on the Mini-EAT survey
Healthy Eating and Weight Self-Efficacy (HEWSE) score | Current self-efficacy at baseline and immediately post-assessment
  The HEWSE is a self-report questionnaire that assesses healthy eating and healthy weight self-efficacy. The scores range from 1-5 with higher scores indicating better self-efficacy.
Motivation for Dietary Self-Control Scale score | Current motivation at baseline and immediately post-assessment
  The Motivation for Dietary Self-Control Scale is a self-report questionnaire that assesses motivations for dietary change with three sub scales: Dietary Goal-Desire Incongruence, Motivation for Dietary Self-control, and Satisfaction with Dietary Behavior. The scores for each subscale range from 0-6 with higher scores indicating better motivation.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Profile v2.0 score | Past 7-day symptoms at baseline and immediately post-assessment
  The PROMIS is a self-report questionnaire measuring overall physical and mental health. PROMIS scores range from 0-5 with higher scores indicating worse mental and physical health.
Body Mass Index value | Current at baseline and immediately post-assessment
  Body mass index is calculated using measured height and weight. Higher scores indicate greater obesity risk.
Hemoglobin A1C (HbA1c) recording | Current at baseline and immediately post-assessment
  HbA1c is calculated using finger prick blood test. Values typically range from 5 to 12 with lower scores indicating less diabetes risk.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler B Mason, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No